CLINICAL TRIAL: NCT04188691
Title: A Randomized, Blind, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Norovirus Bivalent (GI. 1 / GII. 4) Vaccine (Hansenulapolymorpha) in Healthy People Aged 6 Months to 59 Years
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of Norovirus Bivalent Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Lanzhou Institute of Biological Products Co., Ltd (Industry); Beijing Zhong Sheng Heng Yi Pharmaceutical Technology Co., Ltd. (Unknown); Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CXSL1700011-I
Record Dates: First submitted 2019-11-27; First posted 2019-12-06 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2020-04

CONDITIONS: Norwalk Gastroenteritis; Norovirus Infections
MeSH Terms: conditions — Caliciviridae Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- vaccine group 1 (Experimental): vaccine produced by NVSI , Specification: GI.1 / GII.4 (low), 0.5ml / dose
  Interventions: Biological: Norovirus Bivalent (GI.1 / GII.4) Vaccine（low）
- vaccine group 2 (Experimental): vaccine produced by NVSI , Specification: GI.1 / GII.4 (middle), 0.5ml / dose
  Interventions: Biological: Norovirus Bivalent (GI.1 / GII.4) Vaccine（middle）
- vaccine group 3 (Experimental): vaccine produced by NVSI , Specification: GI.1 / GII.4 (high), 0.5ml / dose
  Interventions: Biological: Norovirus Bivalent (GI.1 / GII.4) Vaccine（high）
- Normal saline (Placebo Comparator): （0.5ml / dose）produced by NVSI
  Interventions: Biological: Normal saline
- Aluminum adjuvant (Placebo Comparator): （0.5ml / dose）produced by NVSI
  Interventions: Biological: Aluminum adjuvant

INTERVENTIONS:
Biological: Norovirus Bivalent (GI.1 / GII.4) Vaccine（low） — Norovirus Bivalent (GI.1 / GII.4) Vaccine（low）administered intramuscularly according to a 0, 28，（56） day vaccination schedule
  Arms: vaccine group 1
Biological: Norovirus Bivalent (GI.1 / GII.4) Vaccine（middle） — Norovirus Bivalent (GI.1 / GII.4) Vaccine（middle）administered intramuscularly according to a 0, 28，（56） day vaccination schedule
  Arms: vaccine group 2
Biological: Norovirus Bivalent (GI.1 / GII.4) Vaccine（high） — Norovirus Bivalent (GI.1 / GII.4) Vaccine（high）administered intramuscularly according to a 0, 28，（56）day vaccination schedule
  Arms: vaccine group 3
Biological: Normal saline — Normal saline administered intramuscularly according to a 0, 28 ，（56）day vaccination schedule
  Arms: Normal saline
Biological: Aluminum adjuvant — Aluminum adjuvant administered intramuscularly according to a 0, 28，（56） day vaccination schedule
  Arms: Aluminum adjuvant

SUMMARY:
A total of 450 subjects were enrolled, divided into four age groups, including 18-59 years, 6-17 years, 3-5 years, and 6-35 months. There are three types of the test vaccine component in each age group. A total of 30 people in each dose group were vaccinated with the test vaccine or placebo 1 or placebo 2, respectively, in a ratio of 3: 1: 1.

The 18-59-year-old, 6-17-year-old, and 3-5-year-old age groups were vaccinated 2 times at a time interval of 28 days. The 6-35 month age group is divided into two groups, Group 1 is inoculated with 2 doses interval of 28 days each, and Group 2 is inoculated with 3 doses interval of 28 days.

DETAILED DESCRIPTION:
From January to April 2020, this study was affected by the COVID-19 epidemic, which caused the two groups（6-17-year-old，3-5-year-old） of subjects to vaccinate beyond the window and deviate from the experimental plan. After communication between the researcher, the sponsor and the statistician, it was decided to restart the Phase I clinical trials of these two groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months to 59 years old, can provide legal identification of Chinese population;
* Based on medical history and physical examination, determined by the researcher as healthy;
* Volunteer legal guardians or trustees have the ability to understand (non-illiterate) research procedures, sign informed consent voluntarily with informed consent, and be able to comply with the requirements of clinical research protocols;
* Female subjects of childbearing age were not pregnant at the time of enrollment (negative urine pregnancy test), were not breastfeeding, and had no birth plan within the first 3 months after enrollment; effective contraceptive measures were taken within 2 weeks before enrollment.

Exclusion Criteria:

* Axillary body temperature before inoculation on the day of entry> 37.0 ℃;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc .;
* Have a history of epilepsy, convulsions or convulsions, or a family history of mental illness;
* Those who received immunoenhancement or inhibitor therapy within months (continuous oral or instillation for more than 14 days);
* Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* No spleen or spleen function defect caused by any situation;
* Severe liver and kidney disease, drug-uncontrollable hypertension (systolic blood pressure> 140mmHg, diastolic blood pressure> 90mmHg), diabetic complications, malignant tumors, various acute diseases or chronic attacks of acute diseases;
* Have a history of chronic gastrointestinal diseases, diarrhea or other digestive system diseases, and have had gastroenteritis requiring treatment in the past 7 days;.
* Have a history of abnormal coagulation function (such as coagulation factor deficiency, coagulopathy);
* Have a history of severe allergic reactions to vaccination; are allergic to any component of the test vaccine;
* Live attenuated vaccine within14 days; other vaccines received within 7 days;
* Participating in other clinical trials in the near future;
* The investigator judges other circumstances that are not suitable for participation in this clinical trial.

In addition to the general exclusion criteria, specific populations should also adhere to the following exclusion criteria:

* Premature birth (delivery before the 37th week of pregnancy), low weight (birth <2300g) infants under 24 months of age;
* History of salvage, birth apnea, or other causes of salvage, neurological damage, severe chronic disease (such as Down syndrome, sickle cell anemia, or neurological disorders) in children under 24 months of age.

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 510 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

PRIMARY OUTCOMES:
AE of local and systemic reactions within 30 minutes after each dose | 30 minutes
All active AEs within 0-7 days after each dose | 7 days
  Active AE: Local and systemic adverse reactions occurring within 0-7 days after each dose of vaccination
All non-active collection AEs within 0-28（30） days after each dose | 28（30） days
  Adverse events other than active AE include solicitation adverse events reported in addition to the specified solicitation time window
All SAEs within 6 months after the last dose is vaccinated | 6 months

SECONDARY OUTCOMES:
Calculate geometric mean titer (GMT) of NoV GI.1 and GII.4 IgG antibodies | 28 days after the full vaccination
Calculate positive rate of NoV GI.1 and GII.4 IgG antibodies | 28 days after the full vaccination
Calculate NoV GI.1 and GII.4 HBGA-blocking antibody titers | 28 days after the full vaccination
Calculate NoV GI.1 and GII.4 HBGA-blocking antibody positive rates | 28 days after the full vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- qixian Center for Disease Control and Prevention, Hebi, Henan, China

IPD SHARING:
Plan to Share IPD: No